CLINICAL TRIAL: NCT03843944
Title: Overnight Switch From Rasagiline To Safinamide In Fluctuating Patients With Parkinson's Disease: A Tolerability And Safety Study
Brief Title: Overnight Switch From Rasagiline To Safinamide
Acronym: SWH-MAOB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP 05/17
Record Dates: First submitted 2019-02-12; First posted 2019-02-18 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: IMAO-B; Safinamide; Rasagiline
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safinamide (Experimental): Overnight switch from rasagiline 1 mg OD to safinamide 50 mg OD
  Interventions: Drug: Safinamide

INTERVENTIONS:
Drug: Safinamide — Overnight switch from rasagiline 1 mg OD to safinamide 50 mg OD
  Other Names: Xadago

SUMMARY:
Rasagiline label report the indication to wait at least 14 days between discontinuation of rasagiline and initiation of another MAO inhibitor. This results in a major inconvenience for Parkinsonian patients (PD) due to their clinical worsening. Safinamide is a reversible MAO-B inhibitor, characterized by a good safety profile. In clinical practice safinamide is often introduced instead of rasagiline following an overnight switch. The aim of this study is to explore the safety and tolerability of the immediate switch from rasagiline (irreversible MAO-B inhibitor) to safinamide, with the expectation that there will be no adverse events or increased risk of hypertensive crisis for patients with PD or signs of serotonin syndrome

DETAILED DESCRIPTION:
Objective: The aim of this study is to verify safety and tolerability of the immediate switch from rasagiline to safinamide trough monitoring of BP by 24-hour Holter recording. The primary objective of the study will be achieved if the mean BP will not increase by >10 mmHg in the studied population.

Methods: This is an open-label, single-centre study conducted at IRCCS San Raffaele Pisana. Study population included patients with idiopathic PD in the mid-late stage of the disease, suffering from motor fluctuation, on stable treatment with rasagiline and Levodopa (alone or in combination with other anti-parkinsonian medication). The protocol contemplates five visits during six weeks, with two 24-hour Holter recording (first in rasagiline and second in first-day of safinamide therapy), monitoring typical symptoms of the serotonin syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to comprehend and provide consent form
* Patients with idiopathic Parkinson's disease diagnosed according to the UK Brain Bank criteria
* Patients in mid-to late stage of the disease (Hoehn & Yahr: between the stage 2 and 4 in on state).
* Patients suffering from motor fluctuations
* Patients must have a good response to levodopa in the opinion of the investigators (evaluated as improvement ≥ 30% of the UPDRS scores)
* Stable dosage of antiparkinsonian medication for at least 4 weeks prior to study enrollment
* Female patients in post-menopausal state; women of childbearing potential must use an acceptable method of contraception

Exclusion Criteria:

* Atypical Parkinsonism
* Any significant psychiatric, metabolic and systemic concomitant disease
* Patients with clinically significant out of range laboratory values
* Patients participating in a clinical trial in the last 6 weeks
* Patients with moderate-severe cognitive decline not able to provide consent form
* Patients currently lactating or pregnant or planning to become pregnant during the duration of the study
* Patients for whom Xadago is contraindicated according to the current SmPC

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Blood Pressure (BP) | through study completion, an average of 8 weeks
  Monitoring of BP by 24-hour Holter (increase by >10 mmHg)

SECONDARY OUTCOMES:
Clinical change in UPDRS compared to baseline | through study completion, an average of 8 weeks
  Unified Parkinson's Disease rating scale (UPDRS total score ranges between 0 - normal - to 199 points - severe)
Clinical change in H&Y compared to baseline | through study completion, an average of 8 weeks
  Hoehn and Yahr scale is a system for describing progress of Parkinson's disease (range between 1 -less affect- to 5-more affect)
Clinical change in MoCA compared to baseline | through study completion, an average of 8 weeks
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment (ranges between 0-more affect- and 30-normal)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Stocchi, MD. PhD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Muller T, Hoffmann JA, Dimpfel W, Oehlwein C. Switch from selegiline to rasagiline is beneficial in patients with Parkinson's disease. J Neural Transm (Vienna). 2013 May;120(5):761-5. doi: 10.1007/s00702-012-0927-3. Epub 2012 Nov 30. PMID 23196982
- [Background] Stocchi F, Borgohain R, Onofrj M, Schapira AH, Bhatt M, Lucini V, Giuliani R, Anand R; Study 015 Investigators. A randomized, double-blind, placebo-controlled trial of safinamide as add-on therapy in early Parkinson's disease patients. Mov Disord. 2012 Jan;27(1):106-12. doi: 10.1002/mds.23954. Epub 2011 Sep 12. PMID 21913224
- [Background] Marquet A, Kupas K, Johne A, Astruc B, Patat A, Krosser S, Kovar A. The effect of safinamide, a novel drug for Parkinson's disease, on pressor response to oral tyramine: a randomized, double-blind, clinical trial. Clin Pharmacol Ther. 2012 Oct;92(4):450-7. doi: 10.1038/clpt.2012.128. Epub 2012 Sep 5. PMID 22948897